CLINICAL TRIAL: NCT04599946
Title: Effects of Infant Feeding with Goat Milk Formula or Cow Milk Formula on Atopic Dermatitis
Brief Title: Goat Infant Formula Feeding and Eczema (the GIraFFE Study)
Acronym: GIraFFE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dairy Goat Co-operative (N.Z.) Limited (Industry)
Collaborators: Klinikum der Universität München (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DGC201911
Record Dates: First submitted 2020-10-05; First posted 2020-10-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Dermatitis, Atopic; Eczema, Infantile; Infant Development; Child Development
Keywords: Atopic Dermatitis; Healthy Term Infants; Infant Formula; Infant Development; Child Development
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadrupole
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental formula (Experimental): Infant and follow-on goat milk formula
  Interventions: Dietary Supplement: Infant formula and follow-on formula made from whole goat milk
- Control formula (Active Comparator): Infant and follow-on cow milk formula
  Interventions: Dietary Supplement: Infant formula and follow-on formula made from cow's milk ingredients

INTERVENTIONS:
Dietary Supplement: Infant formula and follow-on formula made from whole goat milk — Infant formula and follow-on formula made from whole goat milk
  Arms: Experimental formula
Dietary Supplement: Infant formula and follow-on formula made from cow's milk ingredients — Infant formula and follow-on formula made from cow's milk ingredients
  Arms: Control formula

SUMMARY:
To determine the relative risk of developing atopic dermatitis in infants fed a study formula based on whole goat milk compared to infants a study formula based on cow milk protein.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, parallel-group trial to study the effect of feeding infants goat milk or cow milk formula in the first year of life on the risk of allergy and other health outcomes, including growth, tolerance and quality of life in the first 5 years of life.

ELIGIBILITY:
Inclusion Criteria:

* Having obtained written informed consent (signed and dated) of the child's parent(s)/caregiver(s), indicating that the child's parent(s)/caregiver(s) has/have been informed of all pertinent aspects of the study
* Born full term (≥37 weeks +0 days and ≤ 41 weeks +6 days of gestation)
* Age at enrolment < 3 months of age (<90 days)
* Birth weight ≥2.5 kg and ≤4.5 kg
* Born from a singleton pregnancy
* Child's parent(s)/caregiver(s) is/are of legal age of consent
* The child's parent(s)/caregiver(s) have sufficient local language skills to understand the study information, the informed consent, and to comply with the study procedure
* The child's parent(s)/caregiver(s) is/are willing and deemed able to fulfil the requirements of the study protocol and procedures
* Mother has expressed the intention to partially (in combination with breastfeeding) or fully formula-feed

Exclusion Criteria:

* Diagnosed disorder considered to interfere with nutrition, growth or development of the immune system
* Participation of the child in any other interventional trial or participation of the mother in any intervention trial with child follow-up
* Infant has a doctor's diagnosis of atopic dermatitis or a severe widespread skin condition prior to randomization that would make the detection or assessment of atopic dermatitis difficult
* Infant has consumed an infant formula for more than 4 weeks prior to enrolment
* Cow milk allergy or intolerance
* Institutionalized infant

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2132 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis up to the age of 12 months | Age 12 months
  Cumulative incidence of atopic dermatitis up to the age of 12 months diagnosed by study personnel (defined as meeting the UK Working Party Diagnostic Criteria for atopic dermatitis)

SECONDARY OUTCOMES:
Cumulative incidence of atopic dermatitis up to the age of 24 and 60 months | Age 24 and 60 months
  Cumulative incidence of atopic dermatitis up to the age of 24 and 60 months diagnosed by study personnel (defined as meeting the UK Working Party Diagnostic Criteria for atopic dermatitis)
Cumulative incidence of parental reported diagnosis of atopic dermatitis up to the age of 12, 24 and 60 months | Age 12, 24 and 60 months
  Cumulative incidence of parental reported diagnosis of atopic dermatitis up to the age of 12, 24 and 60 months, defined as meeting the UK Working Party Diagnostic Criteria for atopic dermatitis
Point incidence of atopic dermatitis | at 4, 6, 12, 24 and 60 months of age
  Point incidence of study and parental diagnosis of atopic dermatitis, defined as meeting the UK Working Party Diagnostic Criteria for atopic dermatitis at the age of 4, 6, 12, 24 and 60 months
Time to onset of atopic dermatitis | Age 12, 24 and 60 months
  Age at first study or reported diagnosis of atopic dermatitis up to the age of 12, 24 and 60 months
Severity of atopic dermatitis | at 4, 6, 12, 24 and 60 months of age
  Atopic dermatitis severity in children with diagnosed (study diagnosis or reported diagnosis) atopic dermatitis, using the SCORing Atopic Dermatitis (SCORAD; Severity Score: 0 to 104, with a higher score indicating more severe eczema) questionnaire completed by a study nurse at all face-to-face visits at 4, 6, 12, 24 and 60 months of age.
Severity of atopic dermatitis | at 4, 6, 8, 10, 12, 18, 24, 36, 48 and 60 months of age
  Atopic dermatitis severity in children with diagnosed (study diagnosis or reported diagnosis) atopic dermatitis, using the Patient Orientated Eczema Measure (POEM; Severity Score: 0 to 28, with a higher score indicating more severe eczema) questionnaire completed by parents at 4, 6, 8, 10, 12, 18, 24, 36, 48 and 60 months of age
Cumulative use of atopic dermatitis-related medication | Age 12, 24 and 60 months of age
  Cumulative use of eczema-related medication or skin care for eczema up to 12, 24 and 60 months of age
Cumulative incidence of atopic dermatitis in risk-related subgroups | Age 12, 24 and 60 months of age
  Cumulative incidence of atopic dermatitis in risk-related subgroups up to 12, 24 and 60 months of age
Incidence of parental reported food allergy | Age 12, 24 and 60 months of age
  Parental report of a clinical diagnosis of food allergy at 12, 24 and 60 months of age
Incidence of allergic sensitization to food or non-food allergens | Age 12 and 60 months of age
  Allergic sensitization at 12 and 60 months of age to any of the common allergens (specific and total IgE)
Incidence of hay fever, asthma and asthma-related diseases | Age 12, 24 and 60 months
  Parental reported hay fever and asthma-related diseases (wheezing and allergic rhinitis) up to 12, 24 and 60 months of age
Biochemical markers: blood markers | at 4, 12 and 60 months of age
  Blood: complete blood count (given numbers of different cells per volume and suitable ratios) at 4, 12 and 60 months of age
Biochemical and metabolic markers: blood markers | at 4, 12 and 60 months of age
  Blood: lipidome and metabolome (including more than 300 compounds reported in µmol/liter) at 4, 12 and 60 months of age
Biochemical and metabolic markers: blood markers | at 4, 12 and 60 months of age
  Blood: inflammation markers (including immunoglobulins and cytokines reported as relative units/liter and ng/ml, respectively) at 4, 12 and 60 months of age
Genetic markers: blood markers | at 12 months of age
  Blood: filaggrin gene at 12 months of age
Gut microbiome profile | at 4, 12 and 60 months of age
  Stool: microbiome
Growth parameters | at baseline, 4, 6, 12, 24 and 60 months of age
  Anthropometry: weight (in kg) at baseline, 4, 6, 12, 24 and 60 months of age
Growth parameters | at baseline, 4, 6, 12, 24 and 60 months of age
  Anthropometry: recumbent length (in cm) at baseline, 4, 6, 12, 24 and standard height (in cm) at 24 and 60 months of age
Growth parameters | at baseline, 4, 6, 12, 24 and 60 months of age
  Anthropometry: BMI (weight and height will be combined to report BMI in kg/cm2) at baseline, 4, 6, 12, 24 and 60 months of age
Growth parameters | at baseline, 4, 6, 12, 24 and 60 months of age
  Anthropometry: weight-for-age, length-for-age and BMI-for-age z-scores (WHO growth standards) at baseline, 4, 6, 12, 24 and 60 months of age
Gastrointestinal symptoms | at 4, 6 and 12 months of age
  Parental report of gastrointestinal symptoms using the Infant Gastrointestinal Symptom Questionnaire (IGSQ; Index Score range from 13 to 65, with higher scores indicating greater gastrointestinal symptom burden) at 4, 6 and 12 months of age
Sleep | at 4, 6 and 12 months of age
  Parental report of sleep using the Brief Infant Sleep Questionnaire (BISQ; data in time: hours and minutes of sleep time) at 4, 6 and 12 months of age
Child's wellbeing | at 4, 12, 24 and 60 months of age
  Parental report of quality of life in children using the Infant Toddler Quality of Life questionnaire™ (ITQOL; infant and parent item scales range from 0 to 100, with a higher score indicating better health) at 4, 12, 24 and 60 months of age
Nutrition | at age 4, 6, 8, 10, 12 and 60 months of age
  Nutrition questionnaire at 4, 6, 8, 10, 12 and 60 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, MD, PhD, Principal Investigator — Dr. von Hauner Children's Hospital, LMU University Hospital Munich
Locations (12):
- Dr. von Hauner Children's Hospital, LMU University Hospital Munich, Munich, Germany
- Poland (4):
  - Wojewodzki Specjalistyczny Szpital Dzieciecy, Olsztyn
  - Karol Jonscher's University Hospital, Poznan
  - Medical College of Rzeszow University, Rzeszów
  - Children's Memorial Health Institute, Warsaw
- Spain (7):
  - Unit of Pediatric Gastroenterology and Nutrition, Torrecardenas University Hospital, Almería
  - EURISTIKOS Excellence Centre for Paediatric Research, University of Granada, Granada
  - Department of Neonatology, Hospital Universitario La Paz, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona
  - INCLIVA Health Research Institute, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Instituto de investigacion Sanitaria de Aragon, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferry JM, Galera-Martinez R, Campoy C, Saenz de Pipaon M, Jarocka-Cyrta E, Walkowiak J, Romanczuk B, Escribano J, Gispert M, Grattarola P, Gruszfeld D, Iglesia I, Grote V, Demmelmair H, Handel U, Gallier S, Koletzko B. Effects of infant feeding with goat milk formula or cow milk formula on atopic dermatitis: protocol of the randomised controlled Goat Infant Formula Feeding and Eczema (GIraFFE) trial. BMJ Open. 2023 Apr 13;13(4):e070533. doi: 10.1136/bmjopen-2022-070533. PMID 37055203